CLINICAL TRIAL: NCT06518057
Title: A Multi-Center Phase 2 Study of Hippocampal Avoidance in Craniospinal Irradiation for Leptomeningeal Metastases From Solid Tumors
Brief Title: Hippocampal Avoidance in Craniospinal Irradiation for the Treatment of Leptomeningeal Metastases From Breast Cancer or Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1124476; NCI-2024-05661 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0020569 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Malignant Neoplasm in the Leptomeninges; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Meningeal Carcinomatosis; Lung Neoplasms | interventions — Specimen Handling; Spinal Puncture; Magnetic Resonance Spectroscopy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Proton or Photon VMAT CSI) (Experimental): Patients undergo proton or photon VMAT CSI with HA over approximately 45 minutes once daily (QD) for 10 days (Monday-Friday) in the absence of unacceptable toxicity. Patients also undergo computed tomography (CT) or positron emission tomography (PET)/CT during screening. Additionally, patients undergo additional CT for radiation planning during screening and magnetic resonance imaging (MRI) throughout the trial. Patients may also undergo lumbar puncture (LP) or alternative methods for cerebral spinal fluid (CSF) collection at the discretion of the treating physician and principal investigator throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Electronic Health Record Review; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Radiation: Proton Beam Craniospinal Irradiation; Other: Survey Administration; Radiation: Volume Modulated Arc Therapy; Procedure: Hippocampal-Avoidance Craniospinal Irradiation

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo CSF sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT and/or CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Other: Electronic Health Record Review — Ancillary studies
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Radiation: Proton Beam Craniospinal Irradiation — Undergo proton CSI
  Other Names: Craniospinal Proton Beam Radiation Therapy; p-CSI; Proton Craniospinal Irradiation; Proton Craniospinal Radiation Therapy
Other: Survey Administration — Ancillary studies
Radiation: Volume Modulated Arc Therapy — Undergo photon VMAT CSI
  Other Names: VMAT; Volumetric Modulated Arc Therapy (procedure)
Procedure: Hippocampal-Avoidance Craniospinal Irradiation — Undergo HA
  Other Names: Hippocampal-sparing Craniospinal Irradiation

SUMMARY:
This phase II clinical trial studies how well craniospinal irradiation (CSI) with hippocampal avoidance, using proton therapy or volumetric modulated arc therapy (VMAT), works in treating patients with breast cancer or non-small cell lung cancer (NSCLC) that has spread from the original (primary) tumor to the cerebrospinal fluid (CSF) and meninges (thin layers of tissue that cover and protect the brain and spinal cord) (leptomeningeal metastases). Radiation therapy is an effective treatment in relieving localized symptoms caused by leptomeningeal metastases. However, the type of radiation therapy typically used does not prevent the spread of leptomeningeal disease. CSI (radiation therapy directed at the brain and spinal cord to kill tumor cells) may be able to target all of the areas of possible leptomeningeal tumor spread. CSI may however result in significant neurological side effects due to radiation damage to a part of the brain called the hippocampus. Hippocampal avoidance (HA) reduces the amount of radiation to the hippocampus. Proton or VMAT CSI with HA may be an effective treatment while reducing neurological side effects for patients with leptomeningeal metastases from breast cancer and NSCLC.

DETAILED DESCRIPTION:
OUTLINE:

Patients undergo proton or photon VMAT CSI with HA over approximately 45 minutes once daily (QD) for 10 days (Monday-Friday) in the absence of unacceptable toxicity. Patients may also undergo computed tomography (CT) or positron emission tomography (PET)/CT during screening. Additionally, patients will undergo additional CT for radiation planning during screening and magnetic resonance imaging (MRI) throughout the trial. Patients may also undergo lumbar puncture (LP) or alternative methods for cerebral spinal fluid (CSF) collection at the discretion of the treating physician and principal investigator throughout the study.

After completion of study treatment, patients are followed up at 3, 6, 9, and 12 months, and then at the time of CNS disease progression, up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer or NSCLC malignancies with leptomeningeal metastases established radiographically and/or through CSF cytology
* Patients who are candidates for radiation therapy for the treatment of leptomeningeal metastases
* Patients ≥ 18 years old
* Karnofsky performance status (KPS) ≥ 60 or Eastern Cooperative Oncology Group (ECOG) ≥ 2
* The patient is able to provide informed consent
* Hemoglobin > 8 g/dL
* Absolute neutrophil count > 1,000/mm
* Platelet count > 100,000/mm
* Participants born female at birth must either be of non-reproductive potential (i.e. post-menopausal by history [≥ 60 years old, or with no menses for > 1 year without an alternative medical cause], OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum /urine pregnancy test within 3 weeks prior to starting radiation therapy (RT)
* Patients with reproductive potential must agree to practice two highly effective contraceptive methods

Exclusion Criteria:

* Patients with multiple, serious major neurologic deficits per physician/investigator assessment including encephalopathy
* Patients with extensive systemic disease and without reasonable systemic treatment options
* Patients who are unable to undergo MRI brain and spine with gadolinium contrast
* Previous radiotherapy to the intended treatment site that precludes developing a treatment plan that respects normal tissue tolerances
* Gross ventricular disease
* Brain metastases within 5 mm of the hippocampal contours not previously treated
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Central nervous system (CNS)-progression free survival (PFS) | Up to 12 months
  PFS is defined as time from craniospinal irradiation (CSI) to CNS disease progression or death. CNS-PFS will be summarized using Kaplan-Meier methodology. Median, 95% confidence interval (CI) and Kaplan-Meier plot will be provided. One-sample log-rank test will be used to test if the median CNS PFS of hippocampal avoidance in CSI for leptomeningeal metastases from breast cancer or non-small cell lung cancer (NSCLC) is significantly larger than the expected median CNS PFS with involved-field radiation therapy (IFRT), i.e., 2.5 months. P-value will be provided.

SECONDARY OUTCOMES:
Number of adverse events associated with hippocampal avoidance craniospinal irradiation (HA-CSI) | Up to 12 months
  The analyses of the adverse events associated with HA-CSI will be descriptive in nature. Summary tables and listings will be provided for all reported adverse events (AEs).
Neurocognitive function assessment | Up to 12 months
  Linear mixed models will be used to examine changes in neurocognitive domain (attention, executive functions, memory) performances from pre-RT baseline to 3, 6, and 12 months. Magnitude of change will be examined at each timepoint using standardized effect sizes (e.g., Cohen's d). For each timepoint, the study investigators will examine the proportion of individuals who demonstrate a reliable change in at least 2 (out of 10) test performances as compared to pre-RT baseline performances.
Overall survival (OS) | Up to 12 months
  Comparison of OS between the study group and the historical cohort will be analyzed using stratified log-rank test. OS will be estimated and visualized using Kaplan-Meier methods.

CONTACTS AND LOCATIONS:
Overall Officials: Lia M. Halasz, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No